CLINICAL TRIAL: NCT01480362
Title: Randomized, Controlled Clinical Trial Evaluating the Efficacy and Clinical Effectiveness of Negative Pressure Wound Therapy for the Treatment of Diabetic Foot Wounds When Compared to Standard Wound Therapy
Brief Title: Treatment Study of Negative Pressure Wound Therapy for Diabetic Foot Wounds
Acronym: DiaFu
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: University of Witten/Herdecke (Other)
Collaborators: Kinetic Concepts, Inc. (Industry); Smith & Nephew Wound Management Inc (Industry)
Responsible Party: Principal Investigator, Doerthe Seidel, Head of division for clinical research at the Institute for Research in Operative Medicine, University of Witten/Herdecke
Allocation: Randomized | Model: Parallel | Masking: Single | Purpose: Treatment
Other Study IDs: UWT_1_GKV; DRKS00003347 (Registry Identifier: German Clinical Trials Register)
Record Dates: First submitted 2011-11-23; First posted 2011-11-28 (Estimated); Last update posted 2020-05-05 (Actual); Status verified 2020-04

CONDITIONS: Foot Ulcer, Diabetic
Keywords: Diabetic foot wound; Amputation wound; Chronic wound
MeSH Terms: conditions — Diabetic Foot | interventions — Negative-Pressure Wound Therapy

STUDY DESIGN:
Who Masked: Outcomes Assessor
Masking Description: Wound photographs are analysed by blinded outcome assessors
Oversight: Data Monitoring Committee: Yes

ARMS (2):
- Negative Pressure Wound Therapy (Experimental): The therapy involves the controlled application of sub-atmospheric pressure to the local wound environment,using a sealed wound dressing connected to a vacuum pump.
  Interventions: Device: Negative Pressure Wound Therapy
- Standard Wound Therapy (Active Comparator): Standard wound therapy according to current evidence-based guideline(basic and advanced methods of wound treatment)
  Interventions: Other: Standard Wound Therapy

INTERVENTIONS:
Device: Negative Pressure Wound Therapy — Used therapy systems:
  KCI. V.A.C. Freedom; Acti V.A.C.; INFO V.A.C. to be used with the V.A.C. Granufoam (black), V.A.C. Granufoam Silver and V.A.C. WhiteFoam Smith & Nephew: Renasys GO and Renasys EZ Plus to be used with the Renassys-F/P and Renassys-G Use of the medical devices and applicable consumption items according to manufacturers guidelines and FDA regulations.
  Other Names: Vacuum assisted closure; Vacuum assisted wound closure
  Arms: Negative Pressure Wound Therapy
Other: Standard Wound Therapy — Standard wound therapy according to current evidence-based guideline(basic and advanced methods of wound treatment)
  Other Names: Standard Conventional Wound Therapy
  Arms: Standard Wound Therapy

SUMMARY:
On behalf of a consortium of 19 health insurance companies the Institute for Research in Operative Medicine as part of the University of Witten / Herdecke gGmbH is planning and conducting a clinical study evaluating the efficacy and effectiveness of negative pressure wound therapy in the treatment of wound healing disorders of the foot, which are caused by diabetes mellitus.

This german multicenter study is due to evaluate whether the negative pressure wound therapy or the control therapy (standard wound therapy following the guidelines) is superior.

Patients will be randomly assigned to the two study arms. Both patients and the treatment staff know about the specific allocation to the negative pressure wound therapy or standard wound therapy arm.

A photo documentation and a computer-based evaluation of the wound images will be performed. This is done centrally by independent examiners, who don't know neither the patient nor the treatment assignment.

It is believed that the application of the negative pressure wound therapy systems compared to standard therapy of diabetic foot wounds will lead more frequent and more rapid to the achievement of complete wound closure and that the use of negative pressure wound therapy is an effective and safe therapy option for the treatment of diabetic foot wounds in inpatient and outpatient care.

Patient´s to be included into the study should have either a chronic diabetic foot wound existing longer than 4 weeks whereas dead tissue components must be completely removed by the doctor or a wound after amputation of foot parts.

The study treatment may have already started in the hospital if applicable. The further wound treatment will be mainly performed within outpatient care. Study Participants will return to the study centre for regular study visits or even for wound treatment.

The comparison of the outcomes of both study arms will give valuable information about the efficacy of negative pressure wound therapy in inpatient as well as outpatient care. These results should be provided until the end of 2016 as a basis for the decision of the Federal Joint Committee to answer the question if the negative pressure wound therapy can be approved as a standard service for reimbursement by health insurance companies.

DETAILED DESCRIPTION:
This study project as part of a European tender has the aim to prove efficacy and effectiveness of negative pressure wound therapy in the management of patients with chronic diabetic foot wounds. The tasks within the study project have been assigned to three contractors / institutions.

On behalf of a consortium of 19 health insurance companies with a central contact consisting of the "AOK-Bundesverband GbR", "Verband der Ersatzkassen e.V." (vdek) and the "Knappschaft" these contractors are responsible for conducting the trial.

The Institute for Research in Operative Medicine (IFOM) as part of the University of Witten / Herdecke gGmbH is responsible for the planning, implementation, analysis and publication of the study.

The Private University of Witten / Herdecke takes over the sponsorship of the study project. The duties and responsibilities of the sponsor are transferred to the staff of the Institute for Research in Operative Medicine of University of Witten / Herdecke. The financial support of the clinical study is provided by the manufacturers of the negative pressure wound therapy systems. The task of payment processing and the contractual provisions is taken over by a management company "Gesundheitsforen Leipzig".

Therapy systems used within the treatment arm of the study will be provided by two manufacturers Kinetic Concepts Incorporated (KCI) and Smith & Nephew Inc. All used treatment systems bear the CE mark and will be used within normal conditions of clinical routine and according to manufacturer's instructions.

This research project is performed because of a decision of the Federal Joint Committee Germany, which states that negative pressure wound therapy can´t be accepted as a standard therapy with full reimbursement by the health insurance companies in Germany. This decision is based on the rapid report and the final report of the Institute for Quality and Efficiency in Health Care, which showed through systematic reviews and meta-analysis of previous study projects that an insufficient state evidence regarding the use of negative pressure wound therapy for the treatment of acute and chronic wounds is existing.

This study evaluates the treatment outcome of the application of a technical medical device, which is based on the principle of negative pressure wound therapy (treatment group 1: Intervention Group) in comparison to standard wound therapy (treatment group 2: Control group) in the treatment of chronic foot wounds after adequate (debridement of avital tissue) wound preparation or amputation wounds resulting from a scheduled amputation below the ankle (talocrural articulation), which are caused in the context of a diabetic foot syndrome.

The clinical trial is designed as a national, multicenter, prospective, randomized controlled superiority study. A blinded evaluation of wound photographs will be performed.

Patients will be randomized 1:1 to the treatment arm: negative pressure wound therapy and the control arm: standard wound therapy.

Patients will be stratified according to assignment to the participating institution (hospital) and by Wagner-Armstrong Stadium.

The inclusion and exclusion criteria are based on the presence of a diagnosis of a diabetic foot wound, the regulatory requirements to the participants in a clinical study and the examination and treatment according to current treatment regulations, evidence-based guidelines and the specifications of the manufacturers of the medical devices.

Only patients meeting all inclusion criteria and no exclusion criterion are allowed to be included into the trial.

The aim of this study is to compare the clinical, safety and economic results of both treatment arms.

The primary endpoints to evaluate the efficacy of negative pressure wound therapy in the treatment of chronic foot wounds caused by a diabetic foot syndrome are both the number of complete wound closure within the maximum treatment period (measured in days) as well as the time until complete wound closure. Complete wound closure should be achieved within the maximum study treatment period of 16 weeks.

In addition, secondary clinical endpoints and safety endpoints, patient-reported outcome endpoints and health economic endpoints are evaluated.

The clinical examination includes parameters that can be used for the analysis of resource use in the inpatient and outpatient care. This includes a comparative analysis of parameters of direct and indirect resource use.

Primarily the perspective of the Statutory Health Insurance is considered. As a secondary perspective the view of society was selected.

Sample size calculation was performed considering results of existing trials, which revealed that a number n = 324 patients must be included in the study in order to carry out the analysis of the primary endpoint "Closure rate".

In due consideration of screening failures, discontinuation of therapy of any cause and losses to Follow-Up a screening of a total of 464 patients must be performed to provide the calculated sample size.The primary efficacy analysis is performed using the intention-to-treat group.

Study results will be provided until the end of 2015 to contribute to the final decision of the Federal Joint Committee Germany regarding the general admission of negative pressure wound therapy as a standard of performance within both medical sectors.

ELIGIBILITY:
Inclusion Criteria:

* Presence of diabetes mellitus
* Presence of a foot wound (chronic wounds; amputation wounds) Wagner stage 2-4
* Existence of the foot wound for at least 4 weeks
* Signed informed consent form
* Patient's eligibility of NPWT in the opinion of the treating physician

Exclusion Criteria:

* Age <18 years
* Non-Compliance
* Pregnancy
* Allergies regarding the release of substances from components of each treatment arm
* Severe anemia, wich was not caused by an infection
* Simultaneous participation of patients in another interventional study / previous participation in the same study
* Use of NPWT systems to the study-related foot lesion within a period of 6 weeks prior to study inclusion
* Presence of necrotic tissue with eschar, which can not be removed
* Untreated osteitis or osteomyelitis
* Not examined / unexplored fistula
* Malignancy of the wound
* Exposed: nerves, blood vessels, anastomotic site
* ambulant NPWT of patients receiving anticoagulants (especially heparinization or marcumar therapy) or with otherwise highly impaired clotting function, which have a risk of circulatory relevant bleeding

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 360 (Actual)
Dates: Start 2011-11; Primary Completion 2015-02 (Actual); Study Completion 2015-04 (Actual)

PRIMARY OUTCOMES:
Number of achieved and confirmed wound closures within the maximum study treatment time | 16 weeks
  Complete wound closure is defined as 100% epithelialization; no need for drainage, no need for supportive therapy or a means of assistance and absence of suture material. Wound closure must sustain at least for a period of 14 days and needs to be confirmed within a separate study visit 14 days after the first diagnosis of wound closure.
Time until wound closure within the maximum study treatment time | 16 weeks
  Complete wound closure is defined as 100% epithelialization; no need for drainage, no need for supportive therapy or a means of assistance and absence of suture material. Wound closure must sustain at least for a period of 14 days and needs to be confirmed within a separate study visit 14 days after the first diagnosis of wound closure.

SECONDARY OUTCOMES:
Time until optimal wound bed preparation | 16 weeks
  Time until optimal preparation of the wound bed for further therapy (granulation of at least 95%)
Time until wound closure within the observation period | 6 months
  Time to reach a complete wound closure within the observation period of 6 months
Recurrences | 6 months
  Recurrences within the observation period of 6 months after complete and confirmed wound closure
Amputations | 16 weeks
  Appearance and dimension of amputations
Wound size | 16 weeks
  Wound size over time
Wound tissue qualities | 16 weeks
  Proportion of wound tissue qualities over time
Number of complete wound closures within the observation period | 6 months
  Number of complete wound closures achieved within the observation period of 6 months
Wound-related pain (Numeric Rating Scale) | 16 weeks
  Patient's pain measured with a numeric Rating scale at each study visit
Quality of Life questionaire (EQ-5D) | 6 months
  EQ-5D at inclusion, end of maximum treatment time or end of therapy, Follow-Up after 6 months
Direct costs | within a maximum treatment time of 16 weeks or until end of therapy
  direct medical resource use and costs: hospitalization, outpatient contact with study centre and other providers, reimbursable drugs, medical sundries, adjuvants, reimbursable services direct non-medical resource use and costs: services, travel costs, expenditure of time for patients, expenditure of time for lay care
Indirect costs | within a maximum treatment time of 16 weeks or until end of therapy
  disability, disability pension, premature death
Serious adverse events | 6 months
  All adverse events that result in death, are life-threatening, require inpatient hospitalization or causes prolongation of existing hospitalization, result in persistent or significant disability/incapacity, are a congenital anomaly/birth defect, or require intervention to prevent permanent impairment or damage.
Adverse Events | 16 weeks
  wound specific and device specific adverse events within the maximum study treatment time

CONTACTS AND LOCATIONS:
Overall Officials: Dörthe Seidel, Principal Investigator — Witten Herdecke University
Locations (42):
- Germany (42):
  - Diabetes Klinik GmbH & Co KG, Bad Mergentheim
  - Evangelisches Krankenhaus, Königin Elisabeth Herzberge gGmbH, Berlin
  - Franziskus-Krankenhaus Berlin, Abteilung für Innere Medizin, Berlin
  - Klinikum Bielefeld, Klinik für Allgemeine und Innere Medizin, Bielefeld
  - Gerhard Rothenaicher, Facharzt für Chirurgie, München Bogenhausen, Bogenhausen
  - Knappschaftskrankenhaus Bottrop Klinik für Gefäßchirurgie, Bottrop
  - Tagesklinik Buchloe, Buchloe
  - Gemeinschaftspraxis Schlotmann - Hochlenert - Zavaleta - Haberstock, Cologne
  - Chirurgische Praxisgemeinschaft am Bayenthalgürtel, Praxis Dr. med. Gerald Engels, Cologne
  - Krankenhaus Porz am Rhein, Klinik für Gefäßchirurgie, Cologne
  - Klinikum Darmstadt, Gefäß- und Endovascularchirurgie, Darmstadt
  - Marienhospital Dortmund-Hombruch, Klinik für Innere Medizin / Diabetologie, Dortmund
  - Klinikum Döbeln, Döbeln
  - Diabetische Schwerpunktpraxis, Duisburg
  - Malteser Krankenhaus - St. Franziskus-Hospital, Medizinische Klinik I, Abt. f. Diabetologie, Flensburg
  - Bürgerhospital, Klinik für Diabetologie und Ernährungsmedizin, Frankfurt
  - Klinikum Frankfurt (Oder), Klinik für Gefäßchirurgie, Frankfurt (Oder)
  - Goethe Universität Frankfurt am Main, Klinik für Gefäß- und Endovascularchirurgie, Frankfurt am Main
  - Weißeritztal-Kliniken GmbH Klinik für Gefäßchirurgie-, vaskuläre und endovaskuläre Chirurgie, Phlebologie, Freital
  - Helfenstein Klinik Geislingen, Allgemein- und Viszeralchirurgie, Geislingen
  - Asklepios Kliniken Harburg, Hamburg
  - ASKLEPIOS Westklinikum Hamburg GmbH, Hamburg
  - Paracelsusklinik am Silbersee, Wundzentrum Hannover, Hannover-Langenhagen
  - Westküstenklinikum Heide, Klinik für Visceral- und Gefäßchirurgie, Heide
  - Städtisches Klinikum Karlsruhe GmbH, Karlsruhe
  - Alexianer Krankenhaus Krefeld GmbH, Klinik für Allgemein-, Visceral- und Thoraxchirurgie, Krefeld
  - St. Remigius Krankenhaus Opladen, Leverkusen
  - Klinikum Ludwigsburg, Klinik für Gefäßchirurgie, vaskuläre und endovaskuläre Chirurgie, Ludwigsburg
  - Diabetologikum Ludwigshafen, Diabetes-Schwerpunktpraxis, Ludwigshafen
  - Uniklinik Lübeck, Klinik für Allgemeine Chirurgie, Lübeck
  - Kliniken Maria Hilf GmbH, Mönchengladbach
  - Städt. Klinikum Bogenhausen, München
  - Institut für Diabetesforschung Münster GmbH, Münster
  - Städtisches Klinikum Neunkirchen gGmbH, Neunkirchen
  - Gemeinschaftspraxis Drs. Alter, Heim, Pourhassan, Oberhausen
  - Ortenau Klinikum Offenburg, Klinik für Allgemein-, Viszeral- und Gefäßchirurgie, Offenburg
  - Klinikum Dorothea Christiane Erxleben Quedlinburg GmbH, Klinik für Allgemein-, Visceral- und Gefäßchirurgie, Quedlinburg
  - Hegau-Bodensee Klinikum Radolfzell (HBK), Klinik für Innere Medizin, Radolfzell
  - Thüringen Kliniken "Georgius Agricola", Klinik für Gefäßchirurgie, Saalfeld
  - St. Marienkrankenhaus Siegen gGmbH, Klinik für Gastroenterologie, Siegen
  - Mariannen-Hospital Werl, Abteilung für Chirurgie, Werl
  - HSK - Dr. Horst Schmidt Kliniken GmbH, Wiesbaden

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Background] Seidel D, Mathes T, Lefering R, Storck M, Lawall H, Neugebauer EA. Negative pressure wound therapy versus standard wound care in chronic diabetic foot wounds: study protocol for a randomized controlled trial. Trials. 2014 Aug 27;15:334. doi: 10.1186/1745-6215-15-334. PMID 25158846
- [Result] Seidel D, Storck M, Lawall H, Wozniak G, Mauckner P, Hochlenert D, Wetzel-Roth W, Sondern K, Hahn M, Rothenaicher G, Kronert T, Zink K, Neugebauer E. Negative pressure wound therapy compared with standard moist wound care on diabetic foot ulcers in real-life clinical practice: results of the German DiaFu-RCT. BMJ Open. 2020 Mar 24;10(3):e026345. doi: 10.1136/bmjopen-2018-026345. PMID 32209619
- [Derived] Seidel D, Lefering R; DiaFu study group. NPWT resource use compared with standard moist wound care in diabetic foot wounds: DiaFu randomized clinical trial results. J Foot Ankle Res. 2022 Sep 30;15(1):72. doi: 10.1186/s13047-022-00569-w. PMID 36180953